CLINICAL TRIAL: NCT02291614
Title: A Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of AMG 211 Administered as Continuous Intravenous Infusion in Subjects With Relapsed/Refractory Gastrointestinal Adenocarcinoma
Brief Title: A Phase 1 Study of AMG 211 in Participants With Advanced Gastrointestinal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated because of immunogenicity and business decision.
Sponsor: Amgen (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20130354; 2014-000201-12 (EudraCT Number)
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: GI Adenocarcinoma
Keywords: Amgen; Phase 1; Clinical Trial; Oncology; GI adenocarcinoma; Immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- AMG 211 200 μg/day for 7/14 Days (Experimental): In cycle 1 participants receive 200 µg/day AMG 211 administered as a continuous intravenous infusion (cIV) infusion at a constant flow rate for 7 days followed by a 3-week treatment-free interval. In cycle 2 and thereafter, participants receive 200 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 200 μg/day for 14 Days (Experimental): Participants receive 200 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 400 μg/day for 14 Days (Experimental): Participants receive 400 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 800 μg/day for 14 Days (Experimental): Participants receive 800 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 1600 μg/day for 14 Days (Experimental): Participants receive 1600 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 1600 µg/day for 28 Days (Experimental): Participants receive 1600 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 3200 µg/day for 14 Days (Experimental): Participants receive 3200 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 3200 µg/day for 28 Days (Experimental): Participants receive 3200 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 6400 µg/day for 14 Days (Experimental): Participants receive 6400 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 6400 µg/day for 28 Days (Experimental): Participants receive 6400 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211
- AMG 211 12,800 µg/day for 28 Days (Experimental): Participants receive 12,800 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
  Interventions: Drug: AMG 211

INTERVENTIONS:
Drug: AMG 211 — continuous intravenous infusion (cIV) infusion in cycles from 7 to 28 days
  Other Names: MEDI-565; MT111

SUMMARY:
The purpose of this Phase 1 study is to determine if AMG 211 given as a continous intravenous (IV) infusion is safe and tolerable in adult participants that have advanced gastrointestinal adenocarcinoma. The study will be conducted in multiple sites and test increasing doses of AMG 211. The safety of participants will be monitored by intensive assessment of vital signs, electrocardiograms, physical examinations, and laboratory tests. Efficacy will be assessed by the usual imaging procedures and their interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided
* 18 years or older
* Advanced relapsed/refracted gastrointestinal adenocarcinoma
* At least 1 measurable tumor lesion
* Tumor tissue available or is willing to undergo biopsy of a tumor lesion before the start of treatment
* Adequate hematological, renal, and liver function
* Body weight ≥ 45 kg
* Other inclusion criteria may apply

Exclusion Criteria:

* Malignancy other than gastrointestinal (GI) adenocarcinoma requiring current therapy
* Evidence of uncontrolled systemic disease, active infection, Hepatitis B and/or C, human immunodeficiency virus (HIV), history of cardiac disease, history of significant central nervous system (CNS) disease, history of chronic autoimmune disease (with the exception of stable type 1 diabetes)
* Major surgery within 28 days of study day 1
* Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment in another investigational device or drug study. Other investigational procedures while participating in this study are excluded. Exception to this criterion is the participation in the optional Imaging Study and all procedures related to this study.
* Treatment with any chemotherapy, radiotherapy, immunotherapy, biologic, or hormonal therapy for cancer within 14 days prior to study entry and not recovered from treatment
* Unresolved toxicities from prior anti-tumor therapy
* Males or Females of reproductive potential, and unwilling to practice an acceptable method of effective birth control while on study through 30 days after receiving the last dose of study drug
* Females who are pregnant, planning to become pregnant, lactating/breastfeeding or who plan to breastfeed while on study through 30 days after receiving the last dose of study drug
* Other exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11-27 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- Germany (3):
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Ulm
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Groningen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in the Netherlands and Germany. Participants were enrolled from 27 November 2014 to 28 March 2017.
Pre-assignment Details: This study was to be conducted in 2 parts: dose-escalation and dose-expansion (planned to enroll additional participants to gain further clinical experience with AMG 211). The dose expansion part was not conducted (study terminated early). In the dose-escalation cohorts, participants were assigned sequentially into cohorts as they opened.
Groups:
- AMG 211 200 µg/Day for 7/14 Days: In cycle 1 participants received 200 µg/day AMG 211 administered as a continuous intravenous (cIV) infusion at a constant flow rate for 7 days followed by a 3-week treatment-free interval. In cycle 2 and thereafter, participants received 200 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- AMG 211 200 µg/Day for 14 Days: Participants received 200 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- AMG 211 400 µg/Day for 14 Days: Participants received 400 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- AMG 211 800 µg/Day for 14 Days: Participants received 800 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- AMG 211 1600 µg/Day for 14 Days: Participants received 1600 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- AMG 211 1600 µg/Day for 28 Days: Participants received 1600 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
- AMG 211 3200 µg/Day for 14 Days: Participants received 3200 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- AMG 211 3200 µg/Day for 28 Days: Participants received 3200 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
- AMG 211 6400 µg/Day for 14 Days: Participants received 6400 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- AMG 211 6400 µg/Day for 28 Days: Participants received 6400 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
- AMG 211 12,800 µg/Day for 28 Days: Participants received 12,800 µg/day AMG 211 administered as a cIV infusion for 28 days followed by a 2-week treatment-free interval.
Period: Overall Study
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Started | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 11 | 2
Received AMG 211 | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2
Completed | 3 | 2 | 2 | 4 | 2 | 2 | 5 | 2 | 3 | 9 | 0
Not Completed | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Decision by sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who enrolled and received at least one dose of study drug.
Groups:
- AMG 211 200 µg/Day for 7/14 Days: In cycle 1 participants received 200 µg/day AMG 211 administered as a cIV infusion at a constant flow rate for 7 days followed by a 3-week treatment-free interval. In cycle 2 and thereafter, participants received 200 µg/day AMG 211 administered as a cIV infusion for 14 days followed by a 2-week treatment-free interval.
- Total: Total of all reporting groups
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days | Total
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.7) | 66.0 (11.5) | 56.7 (12.0) | 60.6 (11.7) | 65.3 (8.1) | 64.0 (4.6) | 64.5 (11.1) | 67.3 (7.6) | 66.0 (13.1) | 62.2 (9.7) | 66.0 (4.2) | 63.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 2 | 0 | 3 | 3 | 1 | 3 | 1 | 21
  Male | 1 | 0 | 1 | 4 | 1 | 3 | 3 | 0 | 2 | 7 | 1 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black (or African American) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 2 | 9 | 2 | 42
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following occurring during the first 28 days of treatment and regarded by the investigator and/or sponsor as related to AMG 211. Hematological DLTs: absolute neutrophil count (ANC) < 0.5 × 10⁹ cells/L for ≥ 7 days; febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection) with ANC < 0.5 × 10⁹ cells/L and fever ≥ 38.5°C; platelets < 25 × 10⁹ cells/L ≥ 7 days. Non-hematological DLTs: any AMG 211-related ≥ grade 3 non-hematological toxicity, excluding nausea and vomiting not refractory to anti-emetics, flare-up of pain due to potential increase in tumor volume, cytokine release syndrome manageable with symptomatic treatment and/or infusion interruption of up to 2 days. The Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 was used to assess toxicities/adverse events.
Time Frame: 28 days
Population: Safety Analysis Set: all participants who enrolled and received at least one dose of AMG 211. Participants were evaluable for a DLT if they received at least 90% of planned doses in the first treatment cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 211 in Cycle 1 in Participants Who Received Dosing for 7 or 14 Days
Description: Levels of AMG 211 in plasma samples collected during this study were analyzed using an electrochemiluminiscence assay. The lower limit of quantification (LLOQ) of the assay was 0.10 ng/mL.
Time Frame: Cycle 1: Predose, 2, 6, 24, 48-96, and 168 (for 14-day dosing groups only) hours after the start of infusion, at the end of infusion (Day 8 or Day 15), and 0.5, 2, 4, 8, and 24 hours after the end of infusion.
Population: Participants who received 7- or 14-day dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 6400 µg/Day for 14 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 3
ng/mL | 5.32 (2.26) [lower limit 2.26] | 11.5 (7.21) [lower limit 7.21] | 13.9 (1.13) [lower limit 1.13] | 19.8 (3.67) [lower limit 3.67] | 55.1 (11.0) [lower limit 11.0] | 116 (32.4) [lower limit 32.4] | 129 (51.0) [lower limit 51.0]

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence, which does not necessarily have a causal relationship with study treatment. A serious adverse event (SAE) was defined as an event that: was fatal or life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/borth defect; or other significant medical event. A TEAE was defined as any AE starting on or after the first dose of study drug and up to and including 30 days after the end of last dose of study drug. The severity of each adverse event was graded using CTCAE version 4.03 criteria (1=mild, 2=moderate, 3=severe, 4=life-threatining, 5=death). 'Any TEAE' includes both serious and non-serious TEAEs.
Time Frame: From first dose of study drug through end of treatment + 30 days (median time frame was 75.5 days).
Population: Safety Analysis Set: all participants who enrolled and received at least one dose of AMG 211.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2
Participants
  Any TEAE | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2
  Grade ≥ 2 TEAE | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 1 | 10 | 2
  Grade ≥ 3 TEAE | 1 | 2 | 2 | 4 | 1 | 2 | 4 | 3 | 1 | 8 | 2
  Grade ≥ 4 TEAE | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0
  Serious TEAE (STEAE) | 1 | 2 | 2 | 4 | 2 | 1 | 6 | 3 | 1 | 9 | 1
  TEAE leading to discontinuation of AMG 211 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0
  STEAE leading to discontinuation of AMG 211 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0
  Non-STEAE leading to discontinuation of AMG 211 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Life-threatening TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Fatal TEAE | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 211 in Cycle 1 in Participants Who Received Dosing for 28 Days
Time Frame: Cycle 1: Predose, 2, 6, 24, 48-96, and 168 hours after the start of infusion, Day 15, at the end of infusion (Day 29), and 0.5, 2, 4, 8, and 24 hours after the end of infusion.
Population: Participants who received 28-day dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 10 | 2
ng/mL | 45.4 (8.86) [lower limit 8.86] | 150 (68.6) [lower limit 68.6] | 145 (45.0) [lower limit 45.0] | 398 (99999) [lower limit 99999]

5. Secondary Outcome: Area Under the Serum Concentration-Time Curve (AUC) From Time 0 to the Last Quantifiable Concentration in Cycle 1 in Participants Who Received Dosing for 7 or 14 Days
Description: Area under the serum concentration-time curve (AUC) from time 0 to the last quantifiable concentration was estimated using the linear trapezoidal method.
Time Frame: as for outcome 2
Population: Participants who received 7- or 14-day dosing.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 6400 µg/Day for 14 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 3
day*ng/mL | 29.7 (19.4) [lower limit 19.4] | 138 (84.7) [lower limit 84.7] | 172 (23.0) [lower limit 23.0] | 214 (77.5) [lower limit 77.5] | 617 (186) [lower limit 186] | 1540 (936) [lower limit 936] | 1420 (666) [lower limit 666]

6. Secondary Outcome: Area Under the Serum Concentration-Time Curve (AUC) From Time 0 to the Last Quantifiable Concentration in Cycle 1 in Participants Who Received Dosing for 28 Days
Description: as for outcome 5
Time Frame: as for outcome 4
Population: Participants who received 28-day dosing.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 10 | 2
day*ng/mL | 1040 (245) [lower limit 245] | 3250 (1700) [lower limit 1700] | 2610 (1940) [lower limit 1940] | 6080 (99999) [lower limit 99999]

7. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Infinity (AUCinf) in Cycle 1 in Participants Who Received Dosing for 7 or 14 Days
Description: Area under the serum concentration-time curve from time 0 to infinity was estimated using the linear trapezoidal method
Time Frame: as for outcome 2
Population: Participants who received 7- or 14-day dosing.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 6400 µg/Day for 14 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 3
day*ng/mL | 30.0 (19.3) [lower limit 19.3] | 140 (85.6) [lower limit 85.6] | 173 (23.4) [lower limit 23.4] | 215 (77.5) [lower limit 77.5] | 619 (186) [lower limit 186] | 1540 (938) [lower limit 938] | 1430 (673) [lower limit 673]

8. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Infinity (AUCinf) in Cycle 1 in Participants Who Received Dosing for 28 Days
Description: Area under the serum concentration-time curve from time 0 to infinity was estimated using the linear trapezoidal method
Time Frame: as for outcome 4
Population: Participants who received 28-day dosing.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 7 | 1
day*ng/mL | 1040 (245) [lower limit 245] | 3260 (1710) [lower limit 1710] | 3180 (2070) [lower limit 2070] | 6530 (99999) [lower limit 99999]

9. Secondary Outcome: Terminal Half-life (T1/2) of AMG-211 in Cycle 1 in Participants Who Received Dosing for 7 or 14 Days
Description: Terminal half-life (t1/2,z) calculated as t1/2,z = ln(2)/λz, where λz was the first-order terminal rate constant estimated via linear regression of the terminal log-linear phase.
Time Frame: as for outcome 2
Population: Participants who received 7- or 14-day dosing.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 6400 µg/Day for 14 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 3
hours | 10.4 (3.34) [lower limit 3.34] | 10.3 (0.703) [lower limit 0.703] | 10.2 (4.37) [lower limit 4.37] | 7.25 (2.63) [lower limit 2.63] | 7.78 (2.37) [lower limit 2.37] | 10.3 (1.72) [lower limit 1.72] | 11.9 (3.53) [lower limit 3.53]

10. Secondary Outcome: Terminal Half-life of AMG-211 in Cycle 1 in Participants Who Received Dosing for 28 Days
Description: as for outcome 9
Time Frame: as for outcome 4
Population: Participants who received 28-day dosing.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 7 | 1
hours | 11.1 (3.45) [lower limit 3.45] | 6.48 (5.16) [lower limit 5.16] | 8.81 (4.58) [lower limit 4.58] | 15.2 (99999) [lower limit 99999]

11. Secondary Outcome: Concentration of AMG 211 at Steady State (Css) in Cycle 1 in Participants Who Received Dosing for 7 or 14 Days
Description: Css was calculated as the average concentration between achievement of plateau and the end of infusion.
Time Frame: as for outcome 2
Population: Participants who received 7- or 14-day dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 6400 µg/Day for 14 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 3
ng/mL | 4.32 (3.27) [lower limit 3.27] | 9.92 (6.05) [lower limit 6.05] | 12.4 (1.73) [lower limit 1.73] | 16.6 (4.42) [lower limit 4.42] | 45.3 (12.9) [lower limit 12.9] | 88.0 (26.4) [lower limit 26.4] | 96.9 (50.8) [lower limit 50.8]

12. Secondary Outcome: Concentration of AMG 211 at Steady State (Css) in Cycle 1 in Participants Who Received Dosing for 28 Days
Description: Css was calculated as the average concentration between achievement of plateau and the end of infusion.
Time Frame: as for outcome 4
Population: Participants who received 28-day dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 10 | 2
ng/mL | 35.9 (7.50) [lower limit 7.50] | 130 (63.9) [lower limit 63.9] | 109 (36.1) [lower limit 36.1] | 306 (99999) [lower limit 99999]

13. Secondary Outcome: Serum Clearance of AMG 211 in Cycle 1 in Participants Who Received Dosing for 7 or 14 Days
Description: Serum clearance (CL) calculated as CL = (actual dose)/(serum concentrations at steady-state [Css] x 24).
Time Frame: as for outcome 2
Population: Participants who received 7- or 14-day dosing.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 6400 µg/Day for 14 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 3
L/hr | 2.93 (2.18) [lower limit 2.18] | 1.36 (1.28) [lower limit 1.28] | 1.36 (0.175) [lower limit 0.175] | 2.13 (0.609) [lower limit 0.609] | 1.57 (0.519) [lower limit 0.519] | 1.62 (0.446) [lower limit 0.446] | 3.21 (1.31) [lower limit 1.31]

14. Secondary Outcome: Serum Clearance of AMG 211 in Cycle 1 in Participants Who Received Dosing for 28 Days
Description: Serum clearance (CL) calculated as CL = (actual dose)/(serum concentrations at steady-state [Css] x 24).
Time Frame: as for outcome 4
Population: Participants who received 28-day dosing.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 10 | 2
L/hr | 1.91 (0.412) [lower limit 0.412] | 1.17 (0.450) [lower limit 0.450] | 2.66 (0.752) [lower limit 0.752] | 1.75 (99999) [lower limit 99999]

15. Secondary Outcome: Volume of Distribution at Steady-state (Vss) in Cycle 1 in Participants Who Received Dosing for 7 or 14 Days
Description: Volume of distribution at steady-state calculated as (CL x t1/2,z)/0.693.
Time Frame: as for outcome 2
Population: Participants who received 7- or 14-day dosing.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 6400 µg/Day for 14 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 3
liters | 50.8 (50.6) [lower limit 50.6] | 20.2 (18.8) [lower limit 18.8] | 19.2 (6.11) [lower limit 6.11] | 22.4 (10.8) [lower limit 10.8] | 18.5 (11.4) [lower limit 11.4] | 23.5 (5.12) [lower limit 5.12] | 50.9 (13.5) [lower limit 13.5]

16. Secondary Outcome: Volume of Distribution at Steady-state (Vss) in Cycle 1 in Participants Who Received Dosing for 28 Days
Description: Volume of distribution at steady-state calculated as (CL x t1/2,z)/0.693.
Time Frame: as for outcome 4
Population: Participants who received 28-day dosing.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 7 | 1
liters | 31.3 (15.0) [lower limit 15.0] | 11.8 (12.4) [lower limit 12.4] | 33.4 (23.5) [lower limit 23.5] | 40.3 (99999) [lower limit 99999]

17. Secondary Outcome: Number of Participants With Anti-AMG 211 Antibody Formation
Description: Blood samples collected during the study were tested for anti-AMG 211 binding antibodies using an electrochemiluminescence-based bridging immunoassay. The number of participants with anti-AMG 211 antibody formation includes participants with a negative or no result at baseline and a positive antibody binding result postbaseline.
Time Frame: Predose and 24 hours after the end of infusion during each treatment cycle, until 4 weeks after the last dose. Median time frame was 75.5 days.
Population: Safety Analysis Set: all participants who enrolled and received at least one dose of AMG 211. Participants with a negative or no result for anti-AMG 211 antibodies at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2
Participants | 1 | 1 | 0 | 3 | 1 | 3 | 5 | 3 | 3 | 10 | 2

18. Secondary Outcome: Number of Participants With an Overall Objective Response
Description: Disease response was assessed by radiological imaging using standardized contrast-enhanced magnetic imaging (MRI) or computed tomography (CT), and evaluated according to the modified Immune-Related Response Criteria (irRC). Overall objective response was defined as a best response of immune-related Complete Response (irCR) or immune-related Partial Response (irPR), confirmed by a repeat, consecutive assessment no less than 4 weeks from the date of the first documented assessment. irCR: Complete disappearance of all lesions and no new lesions. irPR: Decrease in tumor burden ≥ 50% relative to baseline.
Time Frame: Disease response was assessed every second cycle (8-10 weeks) until 4 weeks after the last dose. The median time frame was 75.5 days.
Population: Safety Analysis Set: all participants who enrolled and received at least one dose of AMG 211.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 3 | 3 | 10 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the number of days between the date of the first tumor assessment indicating an objective response through to the subsequent date of progression as classified by modified irRC or death due to any cause. Analyzed in participants with an overall objective response.
  Overall objective response was defined as a best response of immune-related Complete Response (irCR) or immune-related Partial Response (irPR), confirmed by a repeat, consecutive assessment no less than 4 weeks from the date of the first documented assessment. irCR: Complete disappearance of all lesions and no new lesions. irPR: Decrease in tumor burden ≥ 50% relative to baseline.
Time Frame: as for outcome 18
Population: No participant had an objective response.
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Time to Response
Description: Time to response was defined as the number of days from the first administration of AMG 211 to the first objective assessment of response as per modified irRC. Analyzed in participants with an overall objective response.
  Overall objective response was defined as a best response of immune-related Complete Response (irCR) or immune-related Partial Response (irPR), confirmed by a repeat, consecutive assessment no less than 4 weeks from the date of the first documented assessment. irCR: Complete disappearance of all lesions and no new lesions. irPR: Decrease in tumor burden ≥ 50% relative to baseline.
Time Frame: as for outcome 18
Population: No participant had an objective response.
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Time to Tumor Progression in Participants Treated at the Maximum Tolerated Dose (MTD)
Description: Disease was assessed by radiological imaging using standardized contrast-enhanced MRI or CT, and evaluated according to the modified irRC. Immune-related progressed disease (irPD) was defined as an increase in tumor burden ≥ 25% relative to nadir (minimum recorded tumor burden), confirmed by a repeat, consecutive assessment no less than 4 weeks from the date of the first documented assessment.
Time Frame: From first dose of AMG 211 until tumor progression, assessed through the end of study (up to 4 weeks after the last dose). The median time frame was 75.5 days.
Population: Per protocol, only participants treated at the MTD were to be included for this analysis. Because the MTD was not determined in this early-terminated study, this analysis could not be performed.
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Progression Free Survival (PFS) at 6 Months in Participants Treated at the MTD
Description: PFS was defined as the percentage of participants who were progression-free at 6 months.
  Immune-related progressed disease (irPD) was defined as an increase in tumor burden ≥ 25% relative to nadir (minimum recorded tumor burden), confirmed by a repeat, consecutive assessment no less than 4 weeks from the date of the first documented assessment.
Time Frame: 6 months
Population: Per protocol, only participants treated at the MTD for 6 months were to be included for this analysis. Because the MTD was not determined in this early-terminated study, this analysis could not be performed.
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: from enrollment date to end of study date (median time frame was 84 days). Serious and other adverse events: from first dose of study drug through end of treatment + 30 days (median time frame was 75.5 days).
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | AMG 211 200 µg/Day for 7/14 Days | AMG 211 200 µg/Day for 14 Days | AMG 211 400 µg/Day for 14 Days | AMG 211 800 µg/Day for 14 Days | AMG 211 1600 µg/Day for 14 Days | AMG 211 1600 µg/Day for 28 Days | AMG 211 3200 µg/Day for 14 Days | AMG 211 3200 µg/Day for 28 Days | AMG 211 6400 µg/Day for 14 Days | AMG 211 6400 µg/Day for 28 Days | AMG 211 12,800 µg/Day for 28 Days
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/5 | 1/3 | 1/3 | 1/6 | 0/3 | 0/3 | 1/10 | 2/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 2/3 | 4/5 | 2/3 | 1/3 | 6/6 | 3/3 | 1/3 | 9/10 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/5 | 3/3 | 3/3 | 6/6 | 3/3 | 3/3 | 9/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 211 200 µg/Day for 7/14 Days (N=3) | AMG 211 200 µg/Day for 14 Days (N=3) | AMG 211 400 µg/Day for 14 Days (N=3) | AMG 211 800 µg/Day for 14 Days (N=5) | AMG 211 1600 µg/Day for 14 Days (N=3) | AMG 211 1600 µg/Day for 28 Days (N=3) | AMG 211 3200 µg/Day for 14 Days (N=6) | AMG 211 3200 µg/Day for 28 Days (N=3) | AMG 211 6400 µg/Day for 14 Days (N=3) | AMG 211 6400 µg/Day for 28 Days (N=10) | AMG 211 12,800 µg/Day for 28 Days (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hepatic infarction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device infusion issue (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 211 200 µg/Day for 7/14 Days (N=3) | AMG 211 200 µg/Day for 14 Days (N=3) | AMG 211 400 µg/Day for 14 Days (N=3) | AMG 211 800 µg/Day for 14 Days (N=5) | AMG 211 1600 µg/Day for 14 Days (N=3) | AMG 211 1600 µg/Day for 28 Days (N=3) | AMG 211 3200 µg/Day for 14 Days (N=6) | AMG 211 3200 µg/Day for 28 Days (N=3) | AMG 211 6400 µg/Day for 14 Days (N=3) | AMG 211 6400 µg/Day for 28 Days (N=10) | AMG 211 12,800 µg/Day for 28 Days (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 4 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 1 | 1 | 3 | 0 | 0 | 4 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 1 | 0 | 5 | 2
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 3 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Cough decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter removal (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brachiocephalic vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02291614/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02291614/SAP_001.pdf